CLINICAL TRIAL: NCT01452113
Title: Effect of a DPP-IV Inhibitor Treatment on the Secretion of Glucagon in Patients Presenting With Type 1 Diabetes Mellitus With or Without Autonomic Neuropathy
Brief Title: Effect of Autonomic Neuropathy on the Efficacy of a DPP-IV Inhibitor (Galvus) Therapy
Acronym: DPPNAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institute of Molecular Medicine of Rangueil (I2MR) (Unknown); Faculty of Medicine, Toulouse (Unknown); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1004003
Record Dates: First submitted 2011-02-09; First posted 2011-10-14 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; DPP-IV protein; Glucagon-Like Peptide 1; autonomic neuropathy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neuropathy (Other): patients with autonomic neuropathy
  Interventions: Drug: Vildagliptin
- control (Other): patients without autonomic neuropathy (ewing score <= 0.5)
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — one 50 mg tablet per os
  Other Names: GALVUS

SUMMARY:
The purpose of this study is to compare the effect of a single administration of a DPP-IV inhibitor (vildagliptin: Galvus ®) versus no treatment over two populations of diabetic patients: without diabetic autonomic neuropathy (NA, i.e. the control group) and with diabetic autonomic neuropathy (i.e. the neuropathy group). The investigators hypothesize that the therapeutic efficacy of DPP-IV inhibitors is partly mediated by the autonomic nervous system. This hypothesis will be validated if a lower glycemic response to DPP-IV inhibitor treatment is observed for the neuropathy group compared to control.

DETAILED DESCRIPTION:
Recently published work has demonstrated in animals that the control of pancreatic hormone secretion is due, at least in part, to the action of GLP-1 on the via the autonomic nervous system. Therefore, rhe investigators hypothesized that altered autonomic nervous system could explain, at least in part, the altered therapeutic efficacy of DPP-IV inhibitors observed in some patients. Our aim is to validate this concept in humans.

The objective of this physiopathological, monocentric, comparative, open, parallel study is to compare the effect of a single administration of a DPP-IV (vildagliptin: Galvus ®) over two populations of type 1 diabetic patients: a control group of 12 patients without diabetic autonomic neuropathy (NA) and a group of 12 patients with NA.

This proof of concept study will enrol type 1 diabetic patients to avoid confounding factors related to endogen insulin secretion and frequent polymedication of type 2 diabetic patients. The response will be evaluated for each patient by the relative difference between pre-and post-glucagon concentrations following a test meal, measured in the absence and presence of treatment with DPP4 inhibitor. Expected results: the DPP-4 inhibitor should lead to a reduction of about 20 to 30% of the glucagon level in patients without NA and a smaller or no decrease in patients with NA.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* multiple daily insulin injections therapy or continuous insulin infusion (insulin pomp) therapy
* recent (<1 year) written diagnosis of autonomic neuropathy available
* ewing score > 2 for patients to be included in the "neuropathy" group
* ewing score <= 0.5 for patients to be included in the '"control" group
* HbA1C <= 10% at the screening visit and stable (+/- 1%)between the autonomous neuropathy diagnosis and the inclusion visit

Exclusion Criteria:

* severe chronic renal insufficiency defined by an estimated GFR<30 ml/min calculated by MDRD formula)
* proliferative retinopathy needing panphotocoagulation
* hepatic enzymes (ALAT, ASAT) greater than 3 times the upper limit
* congestive heart failure of NYHA functional class III-IV
* clinical signs of gastroparesis
* ongoing gastric emptying therapy
* history of bariatric surgery
* galvus therapy contra indications: known allergy or hypersensitivity of princeps or excipients, galactose intolerance, lapp lactase deficiency, glucose - galactose malabsorption
* ongoing systemic corticoids therapy
* metformin therapy during the day before each study visit
* haemoglobin alteration
* pregnancy or pregnancy willing
* lactation
* ongoing clinical study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
plasma glucagon concentration | 120 min post stantardized meal

SECONDARY OUTCOMES:
GLP-1 | T-30, 0, 15, 30, 60, 90, 120, 180 min post standardized meal
GIP | T-30,0, 15, 30, 60, 90, 120, 180 min post standardized meal

CONTACTS AND LOCATIONS:
Overall Officials: Remy Burcelin, PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Hélène Hanaire, MD PHD, Principal Investigator — UH Toulouse
Locations (1):
- UH Toulouse, Toulouse, France